CLINICAL TRIAL: NCT00672035
Title: Randomized, Double-Blinded, Placebo-Controlled, Dose Ranging Study to Assess the Immunogenicity and Safety of LT Application in Healthy Adults
Brief Title: Prevention, Randomized, Double-Blinded, Placebo-Controlled, Parallel Assignment, Safety/Efficacy Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ELT202
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Traveler's Diarrhea
Keywords: LT; Healthy Adults; Dose Ranging; Patch; Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1 (Experimental): 7.5µg LT Dose placed at the Deltoid on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 2 (Experimental): 7.5µg LT Dose placed at the Lower Back on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 3 (Experimental): 22.5µg LT Dose placed at the Deltoid on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 4 (Experimental): 22.5µg LT Dose placed at the Lower Back on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 5 (Experimental): 37.5µg LT Dose placed at the Deltoid on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 6 (Experimental): 37.5µg LT Dose placed at the Lower Back on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 7 (Experimental): 50µg LT Dose placed at the Deltoid on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 8 (Experimental): 50µg LT Dose placed at the Lower Back on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 9 (Placebo Comparator): Placebo (0µg LT) placed at the Deltoid on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)
- 10 (Placebo Comparator): Placebo (0µg LT) placed at the Lower Back on Day 0 and Day 21
  Interventions: Biological: Biological: heat-labile enterotoxin of E. coli (LT)

INTERVENTIONS:
Biological: Biological: heat-labile enterotoxin of E. coli (LT) — LT patch applied on either the deltoid or the lower back.

SUMMARY:
The main purpose of this study is to evaluate the body's immune response to the LT patch at different doses.

The secondary purpose of this study is to evaluate the safety of the LT patches at different doses and the safety of the skin preparation system. Another secondary purpose is to compare the safety and the body's immune response to LT patches placed on the upper arm versus the lower back.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose ranging, multicenter study. Subjects will be assigned to one of ten treatment groups and vaccinated according to the study group designation. Treatments will remain the same for first and second vaccinations (alternating left and right sides).

ELIGIBILITY:
Subjects must meet all of the following criteria to be eligible to participate in the study:

Inclusion Criteria:

* Healthy adult males or females 18 to 40 years of age with signed informed consent.
* Women who are not post-menopausal or surgically sterile must have a negative serum or urine pregnancy test at screening and within 24 hours prior to each vaccination with understanding (through informed consent process) to not become pregnant over the duration of the study, and must agree to employ an effective form of birth control for the duration of the study.
* Acceptable forms of birth control are: abstinence, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom, diaphragm with spermicide), and IUD.

Subjects meeting any of the following criteria are not eligible for participation in the study:

Exclusion Criteria:

* Laboratory abnormalities.
* Abnormalities at physical examination
* Known allergies to any component of the vaccine.
* Known disturbance of coagulation.
* Known allergies to adhesives.
* Participated in unrelated research involving investigational product within 30 days before planned date of first vaccination.
* Ever received investigational enterotoxigenic E. coli, LT, or LT(R192G) or NasalFlu, Berna Biotech, Ltd.
* Ever received cholera toxin or vaccine (e.g. Orochol™, Dukoral™).
* Medical history of acute or chronic skin disease at vaccination site(s).
* Active skin allergy.
* Recent or regular use of oral or injected steroid medications.
* Use of immunosuppressive systemic steroid medications including inhaled steroids within three months prior to first vaccination.
* Comorbid conditions or treatments that are immunosuppressive, including cancer, diabetes, end-stage renal disease, as determined by the Investigator.
* Positive serology for HIV-1, HIV-2, HBsAg, or HCV.
* History of severe atopy. Signs or history of acute skin infection, sunburn or skin abnormalities on the vaccination area(s) including fungal infections, severe acne, history of keloid formation, or active contact dermatitis.
* Artificial tanning (UV radiation) over the duration of the study including the screening period.
* Hirsute (significant amount of hair) at vaccination area(s).
* Visible tattoos or marks (tattoos/scars) at the vaccination area(s) that would prevent appropriate dermatological monitoring of the vaccination site(s).
* Fever equal to or greater than 38.0°C (≥100.4°F) at the time of planned vaccination.
* Suspicion of or recent history of alcohol or substance abuse.
* Donated blood or blood products such as plasma within the past 30 days.
* Women who are pregnant or breastfeeding.
* Employee of the investigational site.
* Medical history of achlorhydria.
* History of abdominal surgery (excluding C-section, hysterectomy, cosmetic surgery, liposuction, appendectomy, cholecystectomy, ventral hernia repair, and other surgeries not pertaining to gastrointestinal problems) or history of, or recent acute gastrointestinal illness.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 406 (Actual)
Dates: Start 2006-10; Primary Completion 2006-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of LT application at different doses | 6 months

SECONDARY OUTCOMES:
To evaluate the safety of LT application at different doses | 6 months
To evaluate the safety of the skin preparation system | 6 months
To compare patch performance (safety and immunogenicity) on different anatomical parts of the body | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Noss, MD, Principal Investigator — Radiant Research, Cincinnati
Locations (5):
- United States (5):
  - Solano Clinical Research, Davis, California
  - QUEST Research Institute, Bingham Farms, Michigan
  - Asthma and Allergy Associates PC, Cortland, New York
  - Radiant Research - Cincinnati, Cincinnati, Ohio
  - Clinical Trials of Texas, San Antonio, Texas